CLINICAL TRIAL: NCT04543552
Title: A Comparative Analysis of Portable Bladder Scanner to Determine Age/ Volume Specific Accuracy in 0-6 Years of Children
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: H-1709-045-883
Record Dates: First submitted 2020-07-07; First posted 2020-09-10 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2020-07

CONDITIONS: Neurogenic Bladder; Detrusor Underactivity; Detrusor Overactivity
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Urinary Bladder, Underactive; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bladder Scan: Subjects who are scheduled to undergo urodynamic studies.
  Interventions: Device: Bladder scan

INTERVENTIONS:
Device: Bladder scan — Bladder Scanner, or Biocon-900 is an ultrasonic imaging device that has been developed to measure post-void residual volume of the bladder non-invasively. The images and measurements are obtained by applying a probe onto the abdomen (i.e. bladder). As it scans, the scanner constructs 12 cross-sectional images at 15 degree interval using the reflection signals from urine in the bladder and extracts the position of the bladder wall as well. During urodynamic studies, the bladder scan will measure the infused volume in order to assess difference between the infused and scanned volumes.
  Other Names: Bladder Scanner, Biocon-900

SUMMARY:
As a part of the urodynamic studies, urinary catheterization is inserted to measure residual urine, however, it has shown to be an invasive procedure, cause urinary tract infection, and traumatic experience. Bladder scan has been introduced as an alternative and non-invasive method to measure urine residual in the bladder.

DETAILED DESCRIPTION:
Functional urinary disorders are common as more than 15% of children are diagnosed. During the normal course of urinary tract development, bladder and urinary sphincter develop by 2 to 4 years old, and by five years old, the tract is completely developed. The underdevelopment of the urinary tract may lead to complications of the bladder and kidneys along with social impairment. Therefore, the diagnosis is critical as an early diagnosis can prevent long term complications. To diagnose, newborns undergo basic urinalysis, urine culture examination, blood creatinine analysis, and kidney and bladder ultrasound. If any abnormalities are present at the under the age of five, it is recommended that they are followed up on a regular basis. Also, urodynamic studies should be performed every year along with others for early identification and intervention. Studies have shown that UDS (urodynamic studies) significantly reduce the deterioration of the bladder and kidney and the need for operation such as bladder dilation.

As a part of the urodynamic studies, urinary catheterization is inserted to measure residual urine, however, it has shown to be an invasive procedure, which can cause urinary tract infection. The bladder scanner is an ultrasonic imaging device that has been developed for non-invasive measurement of residual volume in the bladder. The images and measurements are obtained by applying a probe onto the abdomen. It constructs 12 cross-sectional images at 15 degree interval using the reflection signals from urine in the bladder and extracts the position of the bladder wall.

The objective of the study is to assess the validity of existing pediatric algorithms for diagnosing neurogenic bladder and evaluate the accuracy of measuring the post-void residual volume between the ages of 0 to 6 years old.

It hypothesizes that when the portable bladder scanner (Bladder Scanner, Biocon-900) is used in pediatric population between the ages of 0 to 3 years old will show greater difference in infused and scanned volume than 4 to 6 years old.

ELIGIBILITY:
Inclusion Criteria:

* Under the age of 6 years old.
* Urodynamic study is scheduled to due to suspected changes in the bladder function or shape.
* Those who understand and sign the informed consent form.

Exclusion Criteria:

* Subjects with surgical history of the bladder.
* Constant leaking of the urine due to bladder neck contracture.
* Any congenital abnormalities that induce changes in the shape of the bladder.
* Unsuitable to participate in the study at the discretion of the principal investigator.

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects who are scheduled to undergo urodynamic studies due to suspected changes in the bladder function or shape.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Scanned bladder volume | Immediately after procedure (urodynamics studies)
  Measurement of the bladder volume
Estimated Post Void Residue | Immediately after procedure (urodynamics studies)
  Estimated PVR
Drainage volume | Immediately after procedure (urodynamics studies)
  Residual urine drained by using a catheter

CONTACTS AND LOCATIONS:
Overall Officials: Kwanjin Park, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No